CLINICAL TRIAL: NCT03006419
Title: Basiliximab vs Reduced Dose Rabbit Antithymocyte Globulin (rRTAG): Evaluation of Efficacy and Safety Outcomes in Low Immunological Risk Living Donor Kidney Transplant: 12-month Randomized Controlled Study
Brief Title: Basiliximab vs Low-dose Thymoglobulin Induction Therapy in Low Risk Kidney Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2016-3001-61
Record Dates: First submitted 2016-12-27; First posted 2016-12-30 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2018-12

CONDITIONS: Kidney Transplant Rejection; Kidney Transplant; Complications
Keywords: kidney transplantation; induction; thymoglobulin; basiliximab; acute rejection; graft loss
MeSH Terms: interventions — Basiliximab; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Basiliximab group) (Active Comparator): Basiliximab (Simulect) induction therapy: 20 mg IV at day of transplant (to be administered 2 hours prior to transplant and up to 4 hours after transplant) and second dosage (20 mg) at fourth day after kidney transplantation.
  Interventions: Drug: Basiliximab
- B (Low-dose Thymoglobulin group) (Experimental): Thymoglobulin induction therapy (1 mg/kg rounded by 25 mg increments) at day of transplant followed by same dosage (1 mg/kg rounded by 25 mg increments) during day 1 and day 2 after transplant in order to complete 3 mg/kg accumulated dose.
  Interventions: Drug: Thymoglobulin

INTERVENTIONS:
Drug: Basiliximab — Standard induction therapy
  Other Names: Simulect
  Arms: Group A (Basiliximab group)
Drug: Thymoglobulin — Induction therapy
  Other Names: rATG
  Arms: B (Low-dose Thymoglobulin group)

SUMMARY:
Demonstrate that low dose (3 mg/kg total ) rATG (thymoglobulin) has similar efficacy (delayed graft function, slow graft function, biopsy proven acute rejection episodes, infections, hospitalizations, adverse events, graft loss and death) than Basiliximab induction

DETAILED DESCRIPTION:
Introduction: The TAILOR study in living donor kidney transplantation demonstrated a 98% one year patient and graft survival and 91% and 83% at 5 years with rejection-free patients in 93%. The cumulative dose of r ATG (thymoglobulin) was 5.29 mg / kg with 3% adverse effects and almost 50% steroid free at 12 months. Others have explored the benefit of low doses of r ATG (thymoglobulin) (3-5 mg / kg) against Basiliximab in low-risk population and demonstrated in living donor recipients with 8 year follow-up similar survival rates with a lower BPAR rate in rATG (thymoglobulin) (p <0.05) and better serum creatinine in 3 and 5 years. The aim of the study was to demonstrate that low dose (3 mg/kg total ) rATG (thymoglobulin) has similar efficacy (delayed graft function, slow graft function, biopsy proven acute rejection episodes, infections, hospitalizations, adverse events, graft loss and death) than Basiliximab induction.

Material and methods: Prospective randomized study of patients undergoing renal transplantation who wish to participate. 100 patients who meet the inclusion and exclusion criteria at the time of transplantation will be randomized

Experimental and reference therapy:

Group A: Induction with Basiliximab 20 mg IV day 0 and day 4 Group B: rATG (Thymoglobulin) 1 mg / kg body weight per day for days 0, 1 and 2 up to a total dose of 3 mg / kg day. According to protocol administration, if there are conditions to delay administration (WBC<2000 / mm3 and / or platelets <75,000 / mm3) (17), administration may be postponed until day 7 posttransplant Posttransplant immunosuppression: Tacrolimus, mycophenolate mofetil and steroids

Outcome measures (12 months) delayed graft function slow graft function biopsy proven acute rejection episodes infections hospitalizations adverse events graft loss death

ELIGIBILITY:
Inclusion Criteria:

* Male or female graft recipients older than 18 years of age.
* Informed consent to participate in the study.
* First living donor kidney transplant recipient.
* Negative pregnancy test if female participant

Exclusion Criteria:

* Second or more kidney transplant.
* Multiple organ transplant recipients.
* ABO incompatibility or positive cross-over test prior to transplantation.
* Antibody Reactive Panel (PRA) > 30%.
* Positive specific donor antibodies (DSA).
* Human immunodeficiency virus (HIV) positive patients.
* HBsAg or HCV positive.
* Severe lung disorders.
* Severe allergies receiving treatment that prevent patient's rRTAG administration.
* Leukocyte count below 2000 / mm3.
* Platelet count below 75,000 / mm3.
* History of malignant disease of any organ system (except skin basal cell carcinoma) within the last 5 years, regardless of local recurrence or metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Biopsy proven acute rejection | 12 months following transplantation
  Acute rejection described by Banff category

SECONDARY OUTCOMES:
Delayed graft function | 12 months following transplantation
  Dialysis during first week of transplantation
Slow graft function | 12 months following transplantation
  Creatinine clearance < 50% pretransplant during first week of transplantation
Infections | 12 months following transplantation
  Presence of a positive culture of any microorganism in presence of clinical symptoms
Hospital admissions | 12 months following transplantation
  Admission to the hospital for at least 24 hours
Graft function | 12 months following transplantation
  Creatinine clearance measured by MDRD-4
Graft loss | 12 months following transplantation
  Return to dialysis
Patient survival | 12 months following transplantation
  Patient Death

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Martinez-Mier, MD, Principal Investigator — Jefe de División, UMAE 189, Veracruz, Veracruz
Locations (1):
- Umae Hospital Especialidades 14 Adolfo Ruiz Cortines, Veracruz, Mexico

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan

REFERENCES:
- [Background] Laftavi MR, Alnimri M, Weber-Shrikant E, Kohli R, Said M, Patel S, Pankewycz O. Low-dose rabbit antithymocyte globulin versus basiliximab induction therapy in low-risk renal transplant recipients: 8-year follow-up. Transplant Proc. 2011 Mar;43(2):458-61. doi: 10.1016/j.transproceed.2011.01.035. PMID 21440733
- [Background] Schenker P, Ozturk A, Vonend O, Kruger B, Jazra M, Wunsch A, Kramer B, Viebahn R. Single-dose thymoglobulin induction in living-donor renal transplantation. Ann Transplant. 2011 Apr-Jun;16(2):50-8. doi: 10.12659/aot.881865. PMID 21716186
- [Result] Brennan DC, Daller JA, Lake KD, Cibrik D, Del Castillo D; Thymoglobulin Induction Study Group. Rabbit antithymocyte globulin versus basiliximab in renal transplantation. N Engl J Med. 2006 Nov 9;355(19):1967-77. doi: 10.1056/NEJMoa060068. PMID 17093248
- [Result] Gaber AO, Matas AJ, Henry ML, Brennan DC, Stevens RB, Kapur S, Ilsley JN, Kistler KD, Cosimi AB; Thymoglobulin Antibody Immunosuppression in Living Donor Recipients Investigators. Antithymocyte globulin induction in living donor renal transplant recipients: final report of the TAILOR registry. Transplantation. 2012 Aug 27;94(4):331-7. doi: 10.1097/TP.0b013e31825a7d1f. PMID 22850297
- [Result] Hardinger KL, Schnitzler MA, Koch MJ, Labile E, Stirnemann PM, Miller B, Enkvetchakul D, Brennan DC. Thymoglobulin induction is safe and effective in live-donor renal transplantation: a single center experience. Transplantation. 2006 May 15;81(9):1285-9. doi: 10.1097/01.tp.0000209825.91632.ea. PMID 16699456